CLINICAL TRIAL: NCT06305182
Title: Metreleptin in Anorexia Nervosa, Randomized Controlled Trial; Effects on Depressive Symptoms and Concomitant Changes in Brain Connectivity
Brief Title: Metreleptin in Anorexia Nervosa
Acronym: METRAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gabriella Milos (Other)
Responsible Party: Sponsor-Investigator, Gabriella Milos, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BASEC 2022-01328
Record Dates: First submitted 2024-02-06; First posted 2024-03-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-05

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Leptin; Metreleptin; Weight gain; Depression
MeSH Terms: conditions — Anorexia Nervosa; Weight Gain; Depression | interventions — metreleptin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized trial. The efficacy of Metreleptin in Anorexia Nervosa patients will be tested against an inactive Placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metreleptin-assisted therapy (Experimental): 25 patients will receive a daily subcutaneous injection of metreleptin for 14 days.
  The dose starts with 0.4 ml daily, and gradually increases until 1.8 ml; until 1.2 ml in male patients daily.
- Placebo-therapy (Placebo Comparator): 25 patients will receive a daily subcutaneous injection of inactive substance (placebo) for 14 days. To ensure blinding, the dosing scheme of placebo will have the identical volume to the dosing scheme of metreleptin (verum).
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Metreleptin — Metreleptin 3 mg is packaged in 3 ml Type I glass vials with chlorobutyl rubber stoppers, and aluminum seals with plastic flip-off caps. The vials are stored in refrigerator (2 - 8°C) and protected from light. Metreleptin for injection is a sterile, white, solid lyophilised cake.
  Prior to patient use, the content of a vial is reconstituted with 0.6 ml of water for injection for a final formulation of 10 millimolar (mM) glutamic acid, 2% glycine, 1% sucrose, 0.01% polysorbate 20, potential hydrogen (pH) 4.25. The resulting solution is administered by subcutaneous injection.
  Other Names: Myalept®
Drug: Sodium chloride — The placebo will consist of sterile 0.9% saline (Sodium chloride), drawn up from a 10 ml i.v. vials. The placebo will be administered as an subcutaneous injection in an identical procedure as the metreleptin verum.
  Arms: Placebo-therapy

SUMMARY:
The treatment of anorexia nervosa often proves to be difficult. There are no drugs that work specifically for the treatment of anorexia nervosa. Experimental administration of metreleptin (synthetically produced leptin) to patients with anorexia nervosa has produced positive results. This study tests the effect of metreleptin in comparison with placebo, which could potentially make treatment easier. The aim of the study is to investigate whether treatment with metreleptin can help to reduce the symptoms of anorexia nervosa and improve mood and weight.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) mainly affects young people, especially young women. AN is one of the most lethal psychiatric disorders. Treatment often proves to be very difficult, and AN course is frequently chronic. Specific pharmacological therapies for AN are lacking. Recent studies have shown that metabolic alterations play a great role in the etiology and pathogenesis of AN. An important metabolic alteration playing a role in the etiology and pathogenesis of AN is the hormone leptin. Patients with AN show hypoleptinemia. The role of hypoleptinemia in the neuroendocrine adaptation to starvation seems to induce emotional, cognitive, and behavioral symptoms of AN. From a theoretical point of view, pharmacotherapy augmenting leptin levels in patients with AN have a great therapeutic potential. Recently, positive effects with experimental administration of subcutaneous metreleptin in few young patients with severe AN have been observed. Importantly, no side effects have been observed. For all these reasons, the present study will investigate - with a double blind design - the therapeutic effect of metreleptin in patients with AN. Metreleptin will be administrated to 50 AN-inpatients: 25 patients will receive verum and 25 will receive placebo during 14 days. Primary objectives of this study are the amelioration of mood and weight. Secondary objectives are the investigation of functional brain connectivity, AN symptoms, as well as hematologic, blood chemistry and neuroendocrinological hormones.

ELIGIBILITY:
Main key inclusion criteria:

* Current diagnosis of AN according to fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) confirmed with Structured Clinical Interview for DSM-5 (SCID-5)
* BMI > 13 kg/m2; BMI ≤ 18 kg/m2; body weight ≥ 35 kg
* Hospitalisation in the Eating Disorders Unit, Department of Consultation-Liaison Psychiatry and Psychosomatic Medicine, University Hospital of Zurich
* Ability to understand German language
* Age range: 17 - 65 years
* Depressive symptoms: HAMD-17 ≥ 8
* Negative urine pregnancy test, non-lactating and double birth control
* Informed Consent as documented by signature

Main key exclusion criteria:

* Illicit drug intake within last month; current alcohol use disorder
* Severe psychiatric and/or severe somatic comorbidities; f. e. lifetime diagnosis of schizophrenia, bipolar disorder, inflammatory bowel disorders, diabetes mellitus, autoimmune disorders, pancreatitis, neurological disorders, cancer including lymphoma
* Acute suicidality or current serious non-suicidal self-injury

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Clinician-rated depression on the 17 point Hamilton Depression Scale (HAMD-17) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  HAMD-17 is a semi-structured interview and consists of 17 items assessing symptoms of depression from the perspective of the clinician. Possible scores range from 0 (no depressive symptom) to 4 (strong depressive symptom). The higher the total score, the more severe the depressive symptoms.
Body weight status in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Body weight status will be indicated by weight in kilograms (kg).

SECONDARY OUTCOMES:
Subjective depression by the Beck Depression Inventory-II (BDI-II) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  The Beck Depression Inventory-II is a self-report rating inventory that measures characteristic attitudes and symptoms of depression with 21 items, ranging from 0 (no depressive symptoms) to 3 (strong depressive symptoms). The higher the total score, the more severe the depressive symptoms.
Functional brain connectivity in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  For assessment of intrinsic functional connectivity in the brain, functional MRI images will be acquired for each patient. A region-of-interest analysis and calculating correlations between any pair of two brain regions, obtaining a connectivity matrix, will be done.
Anorexia Nervosa psychopathology assessed by the Eating Disorders Examination Questionnaire (EDE-Q) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  The Eating Disorders Examination Questionnaire (EDE-Q) is the self-report version of the Eating Disorder Examination (EDE). The 22 items on the four subscales of restraint, eating concern, weight concern, and shape concern are used to assess eating disorder-specific characteristics in their current manifestations during the last 28 days. 7-point rating scales are used to assess frequencies from 0 (characteristic was not present) to 6 (characteristic was present every day or to an extreme degree). Six further, non-scale-forming items also measure the frequency of diagnostically relevant core behaviors over the last 28 days. The EDE-Q is evaluated by calculating subscale mean values for the Restraint, Eating Concern, Weight Concern and Shape Concern subscales and a total score. At Baseline, Post Treatment and intermediate measurements, the instruction of EDE-Q will be modified to refer to a shortened shortened observation time (last week).
External rated hyperkinesia assessed by the Structured Inventory for Anorexic and Bulimic Eating Disorders (SIAB, item 42) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Hyperkinesia will be assessed with only one item (item 42) from the Structured Inventory for Anorexic and Bulimic Eating Disorders (SIAB). This Inventory is used to record the entire spectrum of eating disorder symptoms. Item 42 assesses excessive physical exercise ranging from 0 (no physical exercise) to 4 (very frequent physical exercise).
Subjective hyperkinesia assessed by the Exercise and Eating Disorders Questionnaire (EED) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  The Exercise and Eating Disorders Questionnaire (EED) is a clinically derived, self-report questionnaire. 19 items are used to assess compulsive exercise among eating disorder patients. The 6-point rating scale is used to assess the frequencies (never, rare, sometimes, often, mostly, always) during the last 4 weeks. A higher total score indicates a stronger manifestation of compulsive exercises.
Autism symptoms assessed by the Autism-Spectrum Quotient-short version (AQ-k) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  The Autism-Spectrum Quotient-short version (AQ-k) is a self-assessment tool for screening for autistic disorder. The 10 items represent autistic symptoms and a 4-point response scale is used to assess the agreement (complete agreement, agree more, rather disagree, complete disagreement) to those.
Patient's quality of life by items 1, 2, 5, 6, 7, 10, 17, 19, 20, and 22 from the WHO Quality of Life Questionnaire (WHOQOL-BREF) in the metreleptin-assisted therapy group compared to placebo-therapy between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  The WHO Quality of Life Questionnaire (WHOQOL-BREF) with 26 items is a short form of the WHOQOL-100 and is an instrument for recording subjective quality of life. Items 1, 2, 5, 6, 7, 10, 17, 19, 20, and 22 will be used, ranging from 1 (very dissatisfied/ no agreement) to 5 (very satisfied/fully agreement). A higher total score indicates a increased quality of life.
Visual Analog Scale (VAS) about key Anorexia Nervosa and depression symptoms in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  10 items assessing hunger, repetitive thought of food, fear of weight gain, drive for activity, inner tension, feeling full, nausea, feeling fat, depressed mood and feeling tired on a 10-point response scale ranging from 1 (not pronounced symptom) to 10 (strongly pronounced symptom).
Social interaction by the Liebowitz Social Anxiety Scale (LSAS) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  The Liebowitz Social Anxiety Scale is a clinician-administered assessment that measures the fear and avoidance associated with social anxiety. Item 2,3,4,5,8,10,11,12,15 and 19 will be rated on the response scale for avoidance behavior from 1 (never) to 4 (almost always). Higher scores indicating greater severity of social anxiety.
Anhedonia by the Snaith-Hamilton Pleasure Scale (SHAPS-D) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Anhedonia will be assessed with the german version of the Snaith-Hamilton Pleasure Scale (SHAPS-D) that assesses self-reported anhedonia in psychiatric patients. The respective degree of consent regarding the 14 items on the questionnaire will be rated on a bipolar four-point response scale. For the evaluation, each disagree response ('disagree' or 'strongly disagree') is given 1 point and each agree response is given 0 points. By adding up the points, a higher value indicates a greater degree of anhedonia.
Hematology in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with hemoglobin grams per liter (g/l).
Hematology in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with hematocrit liter per liter (l/l).
Hematology in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with erythrocytes Tera per liter (T/l).
Hematology in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with thrombocytes Giga per liter (G/l).
Hematology in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with leucocytes Giga per liter (G/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with Sodium millimoles per liter (mmol/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with potassium millimoles per liter (mmol/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with phosphate millimoles per liter (mmol/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with creatinine micromoles per liter (µmol/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with creatinine kinase Units per liter (U/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with estimated Glomerular Filtration Rate (eGFR) milliliters per minute (ml/min).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with bilirubin total micromoles per liter (µmol/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with gamma-glutamyltranspeptidase Units per liter (U/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with alanine aminotransferase Units per liter (U/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with alkaline phosphatase Units per liter (U/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with pancreatic amylase Units per liter (U/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with lipase Units per liter (U/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with C-reactive protein (CRP) milligrams per liter (mg/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with calcium millimoles per liter (mmol/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with chloride millimoles per liter (mmol/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with aspartat-aminostransf. (GOT) Units per liter (U/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with magnesium millimoles per liter (mmol/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with protein grams per liter (g/l).
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with albumin grams per liter (g/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with thyroid-stimulating hormon (TSH) milliunits per liter (mU/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with free thyroxin (fT3) picomole per liter (pmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with free thyroxin (fT4) picomole per liter (pmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with follicle stimulating hormone (FSH) international units per liter (IE/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with luteinizing hormone (LH) international units per liter (IE/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with morning cortisol level nanomoles per liter (nmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with fasting insulin millimoles per liter (pmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with leptin nanogram per milliliter (ng/ml).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with ghrelin picogram per milliliter (pg/ml).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with brain derived neurotrophic factor (BDNF) picogram per milliliter (pg/ml).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with cytokine (IL-6) picogram per milliliter (pg/ml).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with cytokine (IL-7) picogram per milliliter (pg/ml).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with estradiol picomole per liter (pmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with testosteron nanomoles per liter (nmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with free testosteron picomole per liter (pmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with progesteron nanomoles per liter (nmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with C-peptide nanomoles per liter (nmol/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with prolactin microgram per liter (µg/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with IGF-1 microgram per liter (µg/l).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with orexin picogram per milliliter (pg/ml).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with oxytocin (unit TBD).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with apodinectin (unit TBD).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with NF-L (unit TBD).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with GFAP (unit TBD).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with leptin receptor (unit TBD).
Neuroendocrinological blood parameters in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with TNF-Alpha (unit TBD).
Heart Frequency Variation (HFV) in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Assessed with ECG and will be analysed with the software HRVTool in Matlab.
Blood chemistry in the metreleptin-assisted therapy group compared to placebo-therapy group between Baseline, Post Treatment and 5 weeks Follow Up | Baseline (day -1), Post Treatment (day 14) and after 5 weeks Follow Up (day 49)
  Measured with Glucose millimoles per liter (mmol/l).

CONTACTS AND LOCATIONS:
Locations (1):
- Eating Disorder Unit, Clinic of Consultation-Liaison Psychiatry and Psychosomatic Medicine, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided